CLINICAL TRIAL: NCT06160115
Title: The Role of Natural Killer Cell Profiling in Predictions of Blood Stream Infection and Antibiotic Resistance in Acute Lymphoblastic Leukemia Patients Post Chemotherapy.
Brief Title: The Role of NK Cells to Detect Blood Infection in ALL.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Sayed Mohamed Ahmed, MSMohamedAhmed, Assiut University
Other Study IDs: NK cells for infection in ALL
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Acute Lymphoblastic Leukemia; Bloodstream Infection
Keywords: Natural Killed cells
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Sepsis | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Flow cytometry — 1. Profiling of NK cells using flow cytometry on peripheral blood and bone marrow aspirate samples.
  2. Isolation and identification of pathogens causing BSI and bacterial drug susceptibility testing using VITEK compact fully automatic microbial identification instrument.
  Other Names: Microbial identification instrument

SUMMARY:
1. Assess possibility of prediction of blood stream infections in ALL patients by profiling of NK cells using flow cytometry.
2. Assess the role of NK cells in development of drug resistance post chemotherapy.

DETAILED DESCRIPTION:
Acute lymphoblastic leukemia (ALL) is the most common malignancy affecting children accounting for approximately 30% of childhood cancers (Zeng XL et al, 2023 ALL is characterized by chromosomal abnormalities and genetic alterations involved in the differentiation and proliferation of lymphoid precursor cells (Fujita, Sousa-Pereira et al. 2021).

ALL is categorized in B-Lymphoblastic Leukemia (B-ALL) And T-Lymphoblastic Leukemia (T-ALL), originated from B- and T-Lineage lymphoid precursor cells, respectively (Chiaretti S et al, 2014).

Recent progress in treatment of ALL has increased the survival rate significantly. The 5-year survival rate in children with ALL is approximately 90% (Paul 2016).

Bloodstream infection is a major cause of treatment-related morbidity and mortality in pediatric patients treated for acute lymphoblastic leukemia (Wolf, Tang et al. 2017).

This is caused by severe and prolonged immunosuppression due to neutropenia, and other chemotherapy-induced alterations of host defense mechanisms The rise of multidrug-resistant bacteria has generated a great challenge to treat infections caused by bacteria with the available antibiotics One of the crucial first line of defense against bloodstream infections in the immune system are Natural Killer cells Natural killer (NK) cells are lymphocytes of the innate immune system that are critical in host defense and immune regulation They can mediate spontaneous cytotoxicity towards malignant cells and microbes, and rapidly secrete numerous cytokines and chemokines to promote subsequent adaptive immune responses

NK cells can be subdivided into different populations based on the relative expression of the surface markers CD16 and CD56

ELIGIBILITY:
Inclusion Criteria:

* Patients aged less than 17 years diagnosed as Acute Lymphoblastic Leukemia and on chemotherapy, who are positive for blood stream infection.

Exclusion Criteria:

1. Patients over 17 years of age.
2. Presence of other hematological malignancies or history of other malignancies.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Primary care clinic.
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who test positive for bloodstream infection and NK cells profile | Baseline
  Assess the number of participants who are positive for bloodstream infection in microbial identification instrument, then comparison of Flow cytometry results for CD16 and CD56 to identify role of NK cells.

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa G Mansour, Professor, Study Chair — South Egypt Cancer Institure, Assiut, Egypt; Eman M Abdel Rahman, Lecturer, Study Chair — Assiut University

REFERENCES:
- [Result] Ammann RA, Laws HJ, Schrey D, Ehlert K, Moser O, Dilloo D, Bode U, Wawer A, Schrauder A, Cario G, Laengler A, Graf N, Furtwangler R, Simon A. Bloodstream infection in paediatric cancer centres--leukaemia and relapsed malignancies are independent risk factors. Eur J Pediatr. 2015 May;174(5):675-86. doi: 10.1007/s00431-015-2525-5. Epub 2015 Mar 26. PMID 25804192
- [Result] Bayatipoor H, Mehdizadeh S, Jafarpour R, Shojaei Z, Pashangzadeh S, Motallebnezhad M. Role of NKT cells in cancer immunotherapy-from bench to bed. Med Oncol. 2022 Dec 2;40(1):29. doi: 10.1007/s12032-022-01888-5. PMID 36460881
- [Result] Bi J, Tian Z. NK Cell Exhaustion. Front Immunol. 2017 Jun 28;8:760. doi: 10.3389/fimmu.2017.00760. eCollection 2017. PMID 28702032
- [Result] Campbell KS, Hasegawa J. Natural killer cell biology: an update and future directions. J Allergy Clin Immunol. 2013 Sep;132(3):536-544. doi: 10.1016/j.jaci.2013.07.006. Epub 2013 Jul 30. PMID 23906377
- [Result] Fujita TC, Sousa-Pereira N, Amarante MK, Watanabe MAE. Acute lymphoid leukemia etiopathogenesis. Mol Biol Rep. 2021 Jan;48(1):817-822. doi: 10.1007/s11033-020-06073-3. Epub 2021 Jan 13. PMID 33438082
- [Result] Gupta DG, Varma N, Naseem S, Sachdeva MUS, Bose P, Binota J, Kumar A, Gupta M, Rana P, Sonam P, Malhotra P, Trehan A, Khadwal A, Varma S. Characterization of Immunophenotypic Aberrancies with Respect to Common Fusion Transcripts in B-Cell Precursor Acute Lymphoblastic Leukemia: A Report of 986 Indian Patients. Turk J Haematol. 2022 Feb 23;39(1):1-12. doi: 10.4274/tjh.galenos.2021.2021.0326. Epub 2021 Oct 7. PMID 34617433
- [Result] Karaman R, Jubeh B, Breijyeh Z. Resistance of Gram-Positive Bacteria to Current Antibacterial Agents and Overcoming Approaches. Molecules. 2020 Jun 23;25(12):2888. doi: 10.3390/molecules25122888. PMID 32586045
- [Result] Littera R, Chessa L, Deidda S, Angioni G, Campagna M, Lai S, Melis M, Cipri S, Firinu D, Santus S, Lai A, Porcella R, Rassu S, Meloni F, Schirru D, Cordeddu W, Kowalik MA, Ragatzu P, Vacca M, Cannas F, Alba F, Carta MG, Del Giacco S, Restivo A, Deidda S, Palimodde A, Congera P, Perra R, Orru G, Pes F, Loi M, Murru C, Urru E, Onali S, Coghe F, Giglio S, Perra A. Natural killer-cell immunoglobulin-like receptors trigger differences in immune response to SARS-CoV-2 infection. PLoS One. 2021 Aug 5;16(8):e0255608. doi: 10.1371/journal.pone.0255608. eCollection 2021. PMID 34352002
- [Result] Lodoen MB, Lanier LL. Natural killer cells as an initial defense against pathogens. Curr Opin Immunol. 2006 Aug;18(4):391-8. doi: 10.1016/j.coi.2006.05.002. Epub 2006 Jun 12. PMID 16765573
- [Result] Matthiesen S, Zaeck L, Franzke K, Jahnke R, Fricke C, Mauermeir M, Finke S, Luhrmann A, Knittler MR. Coxiella burnetii-Infected NK Cells Release Infectious Bacteria by Degranulation. Infect Immun. 2020 Oct 19;88(11):e00172-20. doi: 10.1128/IAI.00172-20. Print 2020 Oct 19. PMID 32817330